CLINICAL TRIAL: NCT03216486
Title: A Phase 2, Non-controlled, Open-Label, Exploratory Study of BPS804 Treatment in Adult Patients With Type I, III or IV Osteogenesis Imperfecta
Brief Title: An Exploratory Study of BPS804 Treatment in Adult Patients With Type I, III or IV Osteogenesis Imperfecta
Acronym: Meteoroid
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative Reason
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBPS208
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — setrusumab

STUDY DESIGN:
Intervention Model Description: Single arm, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BPS804 Dose 1 (Experimental): BPS804 IV Infusion
  Interventions: Drug: BPS804

INTERVENTIONS:
Drug: BPS804 — IV administration of BPS804 in 5% Dextrose solution

SUMMARY:
The purpose of this study is to investigate the effect of BPS804 on strength/quality of bone in patients with Type I, III or IV Osteogenesis imperfecta using a special type of CT scanner. Participants will be treated for 1 year.

DETAILED DESCRIPTION:
This study was previously posted by Mereo Biopharma and was transferred to Ultragenyx in February 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of OI Type I, III or IV
* Capable of giving signed consent

Exclusion Criteria:

* History of skeletal malignancies or other bone diseases (other than OI)
* History of endocrine or thyroid/parathyroid conditions that could affect bone metabolism
* Treatment with bisphosphonates within 3 months of randomisation
* Treatment with teraparatide, denosomab or other anabolic/antiresorbative medications within 6 months of randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-31 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in radial Trabecular Volumetric Bone Mineral Density (mgHA/cm3) | 12 months
  High Resolution Peripheral Quantitative Computated Tomography
Change in radial bone strength on Finite Element Analysis (N) | 12 months
  High Resolution Peripheral Quantitative Computated Tomography

SECONDARY OUTCOMES:
Change in tibial Trabecular Volumetric Bone Mineral Density (mgHA/cm3) | 12 months
  High Resolution Peripheral Quantitative Computated Tomography
Change in tibial bone strength on Finite Element Analysis (N) | 12 months
  High Resolution Peripheral Quantitative Computated Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (2):
- United States (2):
  - Mereo Investigator Site, Albuquerque, New Mexico
  - Mereo Investigator Site, Houston, Texas